CLINICAL TRIAL: NCT01782911
Title: Effect of Resveratrol on Metabolic Parameters and Oocyte Quality in PCOS Patients Undergoing IVF Treatment.
Brief Title: Effect of Resveratrol on Metabolic Parameters and Oocyte Quality in PCOS Patients
Acronym: RES-IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, Medical Doctor, IVI Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAD-IO-01-2013-01
Record Dates: First submitted 2013-01-28; First posted 2013-02-04 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Androgen Profile; Inflammatory Markers; IVF Outcome
Keywords: Androgen; IVF; Resveratrol; PCOS.
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resveratrol (Experimental): Patients will be given 2 g of resveratrol a day from the onset of menses until ovarian pick-up.
  Interventions: Dietary Supplement: Resveratrol
- Control (Placebo Comparator): Patients will be given pills lacking medication from the onset of menses until the ovum pick-up.
  Interventions: Dietary Supplement: Placebo pills

INTERVENTIONS:
Dietary Supplement: Resveratrol — The patients will take 2 g of resveratrol per day for 40 days.
  Arms: Resveratrol
Dietary Supplement: Placebo pills — The patients will take placebo for 40 days.
  Arms: Control

SUMMARY:
Polycystic ovary syndrome (PCOS) is characterized by enlarged ovaries, menstrual irregularity and hyperandrogenism and is the most common cause of oligoovulatory infertility. Insulin resistance with resulting hyperinsulinemia is also common among women with PCOS, along with increased risk for dyslipidemia, hypertension, diabetes and related cardiovascular consequences. Resveratrol is a natural polyphenol with anti-carcinogenic, anti-proliferative and pro-apoptotic properties, that has been shown to decrease proliferation and steroidogenesis in theca cells, emerging as a potential therapeutic agent in PCOS patients. However, little is known about its potential beneficial effect on oocyte quality as well as other reproductive outcomes, such as implantation an pregnancy rates. The present study evaluates effects of resveratrol on selected biochemical parameters and reproductive outcome among patients with PCOS who undergo in vitro fertilization (IVF).

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 18 to 40 years old.
* PCOS diagnosis (according to Rotterdam criteria).
* Mild or moderate male factor, tubal factor or unknown infertility.

Exclusion Criteria:

* Follicle stimulation hormone (third of day of menstruation) > 10 milli international units/L.
* Endometriosis (III o IV).
* Congenital adrenal hyperplasia.
* Cushing syndrome.
* Hyperprolactinemia.
* Thyroid disease.
* Androgenic hormone secretor tumors.
* Patients included in this trial did not take either oral contraceptives, steroids or other medications that could modify the ovarian function, insulin sensitivity or lipid metabolism 3 months before the onset of the trial.
* Severe male factor (sperm concentration < 5 mill/ml).
* Patients undergoing oocyte vitrification to avoid hyperstimulation syndrome will be excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2013-02-01 (Actual); Study Completion 2013-02-01 (Actual)

PRIMARY OUTCOMES:
Effect of resveratrol on oocyte quality | 40 days

SECONDARY OUTCOMES:
Effect of resveratrol on testosterone levels. | 40 days
Effects of resveratrol on inflammatory markers | 40 days
Effects of resveratrol on the fertilization rate. | 40 days
Effects of resveratrol on the pregnancy rate. | 40 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ivi Madrid, Madrid, Spain

REFERENCES:
- [Derived] Showell MG, Mackenzie-Proctor R, Jordan V, Hart RJ. Antioxidants for female subfertility. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007807. doi: 10.1002/14651858.CD007807.pub4. PMID 32851663